CLINICAL TRIAL: NCT00426647
Title: A Randomised Double-blind Multicentre Equivalence Study With Active Parallel Comparator Group to Evaluate the Efficacy and Safety of Norspan® Patches Versus Tramadol in Subjects With Chronic, Moderate to Severe Osteoarthritis Pain in the Hip, Knee &/or Lumbar Spine.
Brief Title: Norspan® Patches Versus Tramadol in Subjects With Chronic, Moderate to Severe Osteoarthritis Pain in the Hip Knee and/or Lumbar Spine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Norpharma A/S (Industry)
Collaborators: Mundipharma Finland (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BUP4006; NORTOP
Record Dates: First submitted 2007-01-23; First posted 2007-01-25 (Estimated); Last update posted 2010-02-01 (Estimated); Status verified 2010-01

CONDITIONS: Osteoarthritis; Pain
Keywords: Osteoarthritis; Pain; Norspan; Buprenorphine; Tramadol
MeSH Terms: conditions — Osteoarthritis; Pain | interventions — Buprenorphine; Tramadol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buprenorphine (Experimental): Norspan transdermal patch
  Interventions: Drug: Buprenorphine
- Tramadol (Active Comparator): Tramadol SR tablets
  Interventions: Drug: Tramadol

INTERVENTIONS:
Drug: Buprenorphine
  Arms: Buprenorphine
Drug: Tramadol
  Arms: Tramadol

SUMMARY:
The primary objective of this equivalence study is to evaluate the efficacy of Norspan® patches versus Tramadol in subjects with chronic, moderate to severe osteoarthritis pain of the hip, knee and/or lumbar spine.

The secondary objectives are to evaluate the safety and general satisfaction for the patients in the two treatment groups.

DETAILED DESCRIPTION:
This is a randomised, double-blind, multicentre equivalence study with active comparator, parallel group, to evaluate the efficacy and safety of Norspan® patches versus Tramadol in subjects with OA pain in hip, knee and/or lumbar spine, currently receiving sub-optimal analgesic treatment (defined as BS-11 score > 4) when treated with paracetamol 4000 mg/day or another analgesic at least comparable to this.

The study consist of 4 phases:

Run-in, Wash-out, Double blind and Follow-up

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18 years or more (women of childbearing potential must have a negative pregnancy test, be non-lactating, and willing to use adequate and reliable contraception (defined as IUD, contraceptive pill or depot gestagen) throughout the study) with osteoarthritis in the hip &/or knee.

   Or Males & females aged 50 years or more with osteoarthritis in lumbar spine without nerve root pressure.
2. Clinical diagnosis of OA in the hip and/or knee including fulfilment of ACR-criteria and radiographic or MR-Scan evidence for the primary OA-joint in hip &/or knee.

   Or Clinical diagnosis of OA in the lumbar spine without nerve root pressure, & with radiographic or CT-scan evidence for lumbar OA.
3. Subjects with moderate to severe pain confirmed by a BS-11 score > 4 for their pain on average in their primary OA-joint during the last 5 days prior to the Baseline Visit (Randomisation Visit/Visit 4).
4. Subjects must previously or during Wash-out-Phase have been treated with 4000 mg Paracetamol IR daily or another analgesic treatment at least comparable to this and not have been adequately pain relieved (defined as BS-11 score > 4 for their pain on average in their Primary OA-joint during 5 continuous days) on that treatment.
5. Subjects must be willing to discontinue all other analgesics (incl. glucosamine) at the Pre-Screening Visit (Visit 1) and until the Completion/Discontinuation Visit (Visit 10).
6. Subjects must be able to read and comprehend Danish and be willing to sign informed consent.
7. Subjects must be willing and able to fill in a Subject Diary on a daily basis.

Exclusion Criteria:

1. Subjects treated with high-potent opioid analgesics (e.g. morphine, fentanyl, oxycodone, methadone, hydromorphone, ketobemidone, buprenorphine (incl. Norspan® patches)) for their OA pain. Except subjects treated with high-potent opioid analgesics for up to four continuous weeks for their OA pain beyond 3 months prior to the Pre-screening Visit.
2. Subjects treated with high-potent opioid analgesics (e.g. morphine, fentanyl, oxycodone, methadone, hydromorphone, ketobemidone, buprenorphine (incl. Norspan® patches)) within four weeks prior to the Pre-screening Visit due to non-OA pain.
3. Subjects treated with more than 200 mg Tramadol daily or 200 mg codeine daily during the last two weeks prior to the Pre-screening Visit.
4. History of chronic condition(s), in addition to OA, requiring frequent analgesic therapy (e.g. frequent headaches, frequent migraine, gout, rheumatoid arthritis) and severe respiratory disease.
5. Scheduled for surgery that would fall within all phases (Run-in-Phase, Wash-out-Phase, Double-Blind-Phase and Follow-up-Phase) of the study.
6. Substance or alcohol abuse, or subjects who, in the opinion of the Investigator, have demonstrated addictive or substance abuse behaviour.
7. Subjects with cancer (except basal cell carcinoma) or history of cancer in the last 5 years (except treated basal cell carcinoma).
8. Untreated depression or other psychiatric disorder in such a way that participation in the study may, in the opinion of the Investigator, pose an unacceptable risk to the subject.
9. Dermatological disorder at any relevant patch application site that precludes proper placement and/or rotation of patch placement.
10. Treatment with steroids (oral, intra-muscular, intra-venous, intra-articular, epidural, or other corticosteroid injections) within 6 weeks prior to the Pre-screening Visit and during the study.
11. Intra-articular hyaluron acid injections given within 6 months prior to the Pre-screening Visit and during the study.
12. Any joint evacuation carried out within 6 weeks prior to the Pre-screening Visit and during the study.
13. Subjects who are currently taking monoamine oxidase inhibitors (MAOIs) or have taken MAOIs within 2 weeks prior to the Pre-screening Visit.
14. Participation in a clinical research study involving a new chemical entity within 3 months prior to the Pre-screening Visit.
15. Allergies or other contraindications to transdermal systems or patch adhesives.
16. Known lack of tolerance and/or effect of Tramadol.
17. Known hypersensitivity (allergic reaction) to opioids or Paracetamol.
18. Ongoing requirement for and treatment with direct external heat sources such as heat lamps, electric blankets, saunas, heating pads and heated waterbeds.
19. New physiotherapy and/or chiropractic and/or other non pharmacological regimen scheduled to commence during the Run-in-Phase, Wash-out-Phase or Double-Blind-Phase of the study. This includes physiotherapy and/or chiropractic and/or other non pharmacological regimen not in a scheduled weekly window.
20. Subjects who cannot or will not cut the hair at the patch site for proper placement of the patch.
21. Any other contraindications listed in the Summary of Product Characteristics for Norspan® patches or Tramadol.
22. Subjects, who are unsuitable for any other reason to participate in the study in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-02; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Equivalence study to evaluate the efficacy of Norspan® patches versus Tramadol in subjects with chronic, moderate to severe osteoarthritis pain of the hip, knee and/or lumber spine.

SECONDARY OUTCOMES:
To evaluate the safety and general satisfaction for the patients in the two treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Dorthe Tvinnemose, DVM, Study Director — Norpharma A/S, Slotsmarken 15, DK-2970 Hoersholm, Denmark; Kim H Kristiansen, DM, Principal Investigator — GP, Noerretorv 10, DK-7200 Grindsted, Denmark; Olavi Airaksinen, DM, Principal Investigator — Oma Lääkäri Oy, Vuorikatu 20, FIN-70100 KUOPIO
Locations (1):
- Dr. Olavi Airaksinen, Oma Lääkäri Oy, Vuorikatu 20, Kuopio, Finland